CLINICAL TRIAL: NCT02236962
Title: Enhancement of Brown Adipose Tissue Function Via Chronic Pharmacological Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bayside Health (Other Government)
Collaborators: Baker Heart and Diabetes Institute (Other); The Alfred (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 15-12
Record Dates: First submitted 2012-01-30; First posted 2014-09-11 (Estimated); Last update posted 2014-09-11 (Estimated); Status verified 2014-09

CONDITIONS: Type 2 Diabetes; Obesity; Cardiovascular Disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Cardiovascular Diseases | interventions — Ephedrine; Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): lactose powder in equivalent capsule
  Interventions: Drug: Placebo
- Drug treatment (Experimental): sympathetic agonist and thiazolidinedione
  Interventions: Drug: Ephedrine, pioglitazone

INTERVENTIONS:
Drug: Placebo
  Arms: Placebo
Drug: Ephedrine, pioglitazone
  Arms: Drug treatment

SUMMARY:
Obesity is epidemic in Australia, and current preventative strategies have had limited success in alleviating this health crisis. While numerous options are available for treatment of obesity, most do not result in sustained weight reduction. Obesity results from an imbalance between energy intake and expenditure, therefore new methods that correct this imbalance are essential for effective long-term treatment. Rodent studies show that brown adipose tissue (BAT) can burn more energy than any other tissue in the body, therefore targeting BAT to increase its activity (energy burning rate) and quantity in humans is potentially a powerful tool for the treatment of obesity and related diseases. BAT has only recently been irrefutably identified in adult humans therefore little is known about how it functions in humans.

ELIGIBILITY:
Inclusion Criteria:

* Males aged 19 - 35 years
* Free of overt coronary disease (on history, medical examination and ECG)
* Unmedicated
* No major illness
* BMI <27 kg/m2

Exclusion Criteria:

* Unable to give informed consent
* Smokers
* Participant in research projects involving ionising radiation within the past 5 years.
* Claustrophobia
* Fasting plasma glucose > 6.0 mmol/L

Ages: 19 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2012-04; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
brown adipose tissue activity | 3 years
  measured via PET-CT

CONTACTS AND LOCATIONS:
Locations (1):
- Alfred Hospital, Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Loh RKC, Formosa MF, Eikelis N, Bertovic DA, Anderson MJ, Barwood SA, Nanayakkara S, Cohen ND, La Gerche A, Reutens AT, Yap KS, Barber TW, Lambert GW, Cherk MH, Duffy SJ, Kingwell BA, Carey AL. Pioglitazone reduces cold-induced brown fat glucose uptake despite induction of browning in cultured human adipocytes: a randomised, controlled trial in humans. Diabetologia. 2018 Jan;61(1):220-230. doi: 10.1007/s00125-017-4479-9. Epub 2017 Oct 18. PMID 29046921
- [Derived] Carey AL, Pajtak R, Formosa MF, Van Every B, Bertovic DA, Anderson MJ, Eikelis N, Lambert GW, Kalff V, Duffy SJ, Cherk MH, Kingwell BA. Chronic ephedrine administration decreases brown adipose tissue activity in a randomised controlled human trial: implications for obesity. Diabetologia. 2015 May;58(5):1045-54. doi: 10.1007/s00125-015-3543-6. Epub 2015 Mar 1. PMID 25725625